CLINICAL TRIAL: NCT05228444
Title: Managing Sleep-wake Disruption Due to Hospitalisation: the Circadian Care Project
Acronym: CircadianCare
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Padova (Other)
Responsible Party: Principal Investigator, Prof.ssa Sara Montagnese, Professor, University Hospital Padova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 150949
Record Dates: First submitted 2022-01-10; First posted 2022-02-08 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Circadian Rhythm Disorders
MeSH Terms: conditions — Chronobiology Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Circadiancare (Experimental): limits the circadian impact of hospitalisation by enhancing circadian rhythmicity through an assessment of the patient's specific circadian features/needs and an ad hoc, personalized light-dark, meal and activity schedule to cover the whole of the inpatient stay.
  Interventions: Behavioral: CircadianCare
- Control (No Intervention)

INTERVENTIONS:
Behavioral: CircadianCare — enhancing circadian rhythmicity through an assessment of the patient's specific circadian features/needs and an ad hoc, personalized light-dark, meal and activity schedule to cover the whole of the inpatient stay.
  Arms: Circadiancare

SUMMARY:
Sleep is regulated by the interaction of homeostatic and circadian processes. The homeostatic process determines sleep propensity in relation to sleep-wake history, the circadian one is responsible for the alternation of high/low sleep propensity in relation to dark/light cues, and is substantially independent of preceding sleep-wake behaviour. The circadian timing system encompasses a master clock in the brain and peripheral, ancillary time-keepers in virtually every organ of the body.

In recent years, evidence has emerged that circadian disruption has serious medical consequences, including sleep loss, increased cardiovascular morbidity and increased risk of certain types of cancer. Evidence is also emerging that hospitalization per se weakens circadian rhythmicity, due to disease itself and to modified light, food and activity cues.

The aim of our project is to test an inpatient management system (CircadianCare) that limits the circadian impact of hospitalisation by enhancing circadian rhythmicity through an assessment of the patient's specific circadian features/needs and an ad hoc, personalized light-dark, meal and activity schedule to cover the whole of the inpatient stay. This will be compared to standard inpatient management in terms of patients' perception, sleep-wake quality and timing during hospitalisation, inpatient utilization of sleep-inducing medication, length of hospitalisation, and prognosis (i.e. outcome of hospitalisation, subsequent hospitalisations and post-discharge sleep-wake disturbances).

The CircadianCare system is expected to benefit prognosis, decrease costs, and change the way hospitals are organized and designed in future, with potential direct relevance to the plans for the new University Hospital of Padova.

ELIGIBILITY:
Inclusion Criteria:

• Hospitalized patients

Exclusion Criteria:

• absence of compliance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-28 (Actual); Primary Completion 2023-01-28 (Estimated); Study Completion 2023-01-28 (Estimated)

PRIMARY OUTCOMES:
Change in sleep onset latency - actigraphy | first, 7th and 14 day
  Sleep latency (number of minutes between try to sleep and sleep onset, SL) is objectively assessed by wrist actigraphy device. SL > 30 min is considered clinically significant. (scale minutes)
Change in sleep onset latency - sleep diary | first, 7th and 14 day
  The number of minutes between try to sleep and sleep onset as measured by sleep diary. Sleep latency > 30 min is considered clinically significant. (scale minutes)
Change in sleep duration - actigraphy | first, 7th and 14 day
  Total sleep time (TST) is calculated as hours per night spent sleeping while in bed after light off. It is objectively assessed by wrist actigraphy device. (scale hours)
Change in sleep duration - sleep diary | first, 7th and 14 day
  Total sleep time (TST) is calculated as hours per night spent sleeping while in bed after light off. It is assessed using daily sleep diaries. (scale hours)
Change in sleep awakening - actigraphy | first, 7th and 14 day
  Measured with wrist actigraphy, wake after sleep onset (WASO) is the number of minutes scored as wake from sleep onset until the end of the last sleep episode while in bed. (scale minutes)
Change in sleep awakening - sleep diary | first, 7th and 14 day
  Measured with sleep diary. Wake after sleep onset (WASO) is a subjective measure of participants' sleeping and waking times in which time awake expressed in minutes after sleep onset is obtained.
Change in sleep efficiency - actigraphy | first, 7th and 14 day
  Measured with wrist actigraphy, sleep efficiency (SE) is the percentage of time (0%-100%) the participant was sleeping from sleep onset (defined as the first 20 continuous minutes of sleep after getting into bed) until the last minute scored as sleep (the following morning).
Change in sleep efficiency - sleep diary | first, 7th and 14 day
  Measured with sleep diary. The sleep efficiency is a subjective measure of participants' sleeping and waking times, from which sleep efficiency is computed as the quota between time sleeping/time spent in bed, expressed in percentage.
Actigraphy - change in fragmentation of activity-rest periods | 14 days
  Interdaily variability (IV) quantifies the degree of fragmentation. The variable has a theoretical range of 0 to 2 with higher values indicating higher fragmentation. Typical values for healthy subjects will be below 1.
Actigraphy - change in sleep regularity over days | 14 days
  Intradaily stability (IS) quantifies the degree of regularity in the activity-rest pattern with a range of 0 to 1 where a value of 0 indicates a total lack of rhythm and a value of 1 indicates a perfectly stable rhythm.
Change in daytime sleepiness | first day then again at 7th and 14th day
  Karolinska Sleepiness Scale (KSS) comprises a single item assessing state sleepiness at a particular time (every hour) during the day on a scale from 1 (very rested) to 9 (very sleepy).
Salivary melatonin shift | baseline DLMO and then again at 7th and 14th day
  A change in the timing of the circadian system is measured using the Dim Light Melatonin Onset (DLMO), gold standard for measuring human circadian phase. Salivary melatonin is measured five times every 1h before usual bedtime and assayed using standard commercially-available radioimmunoassay (RIA) kits. The time at which melatonin rises above a 4 pg/mL threshold is the DLMO.
Diurnal preference | first day
  Short version Munich Chronotype Questionnaire (microMCTQ), measure chronotype based on the midpoint of sleep.
Assess circadian preference | first day
  Morning-evening questionnaire (MEQ) scale: MEQ sum score, range: 16-86, participants are classified as Morning-types (scores between 59 and 86), Neither-types (scores between 42 and 58), and Evening-types (scores between 16 and 41).
Sleep quality | first day
  Pittsburgh Sleep Quality Index (PSQI) scale: global PSQI score, range: 0 - 21, scores of 5 or higher indicate poor sleep quality.

SECONDARY OUTCOMES:
Monitoring environment temperature | first, 7th 14th day
  Temperature levels within ward rooms will be monitored at regular intervals by ibutton temperature sensors, using the Celsius scale.
Monitoring environment noise | first, 7th 14th day
  Noise levels within ward rooms will be monitored at regular intervals by phonometers. Noise level is measured in decibels (dB)

CONTACTS AND LOCATIONS:
Locations (1):
- Padova University Hospital, Padua, Italy

IPD SHARING:
Plan to Share IPD: No